CLINICAL TRIAL: NCT00957723
Title: A Post-market, Non-randomized, Historical Controlled, Multi-center Study of the Outcomes of the Triathlon® Cruciate Retaining (CR) Total Knee System
Brief Title: Triathlon® Cruciate Retaining (CR) Total Knee System Outcomes Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 56
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triathlon® CR Total Knee System (Other): Participants receive the Triathlon® CR Total Knee System
  Interventions: Device: Triathlon® CR Total Knee System

INTERVENTIONS:
Device: Triathlon® CR Total Knee System — The purpose is to evaluate the Triathlon® CR Total Knee System.

SUMMARY:
The purpose of this study is to evaluate the clinical outcomes (range of motion, pain, function, radiographic stability, and health related quality of life) of patients receiving the Triathlon® Cruciate Retaining (CR) Total Knee System. These outcomes will be evaluated by comparing pre-operative to post-operative scores, as well as to a control group. The control group is the Scorpio® CR Total Knee System.

DETAILED DESCRIPTION:
The Triathlon® Cruciate Retaining (CR) Total Knee System components are for use in cemented total knee arthroplasty for painful, disabling joint disease of the knee resulting from non-inflammatory degenerative joint disease (including osteoarthritis, traumatic arthritis or avascular necrosis) or rheumatoid arthritis (excluded from this study according to protocol). The components are designed to improve range of motion (ROM) and stability. This study serves to demonstrate that subjects have reduced pain, increased ROM and improved stability following implantation with the Triathlon Cruciate Retaining (CR) Total Knee System as compared to the historical control.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is a male or non-pregnant female between the ages of 21 and 80.
2. The subject requires a primary cemented total knee replacement.
3. The subject has a diagnosis of osteoarthritis (OA), traumatic arthritis (TA), or avascular necrosis (AVN).
4. The subject has intact collateral ligaments.
5. The subject has signed the IRB-approved, study specific Informed Patient Consent Form.
6. The subject is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

1. Patient has inflammatory arthritis.
2. The subject is morbidly obese, BMI > 40.
3. The subject has a history of total or unicompartmental reconstruction of the affected joint.
4. Patient has had a high tibial osteotomy or femoral osteotomy.
5. The subject has no obvious charcot (i.e. a neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device).
6. The patient has a systemic or metabolic disorder leading to progressive bone deterioration.
7. The subject is immunologically suppressed, or receiving chronic steroids (> 30 days duration).
8. The subject's bone stock is compromised by disease or infection, which cannot provide adequate support and/or fixation to the prothesis.
9. The subject has had a knee fusion to the affected joint.
10. The subject has an active or suspected latent infection in or about the knee joint.
11. The subject is a prisoner.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2005-02; Primary Completion 2010-04 (Actual); Study Completion 2017-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Knute Buehler, MD, Principal Investigator — The Center: Orthopaedic & Neurosurgical Care & Research; Brian Covino, MD, Principal Investigator — Knoxville Orthopedic Clinic; Joseph Davies, MD, Principal Investigator — Aurora Advanced Healthcare; Kenneth Greene, MD, Study Chair — Crystal Clinic; Anthony Hedley, MD, Principal Investigator — Arizona Institute for Bone and Joint Disorders; Kirby Hitt, MD, Principal Investigator — Scott & White Memorial Hospital; Joseph McCarthy, MD, Principal Investigator — Newton-Wellesley Hospital; Jeffrey Nassif, MD, Principal Investigator — Physician's Clinic of Iowa, PC; Kenneth Krackow, MD, Principal Investigator — Buffalo General Hospital, Department of Orthopaedics; Sean Scully, MD, Principal Investigator — Cedars Medical Center University of Miami; Carlton Savory, MD, Principal Investigator — Hughston Sports Medicine Center; Mathew Phillips, MD, Principal Investigator — Buffalo General Hospital, Department of Orthopaedics
Locations (11):
- United States (11):
  - Arizona Institute for Bone and Joint Disorders, Phoenix, Arizona
  - Cedars Medical Center University of Miami, Miami, Florida
  - Hughston Sports Medicine Center, Columbus, Georgia
  - Physician's Clinic of Iowa, Mercy Medical Center, Cedar Rapids, Iowa
  - Newton Wellesley Hospital, Newton, Massachusetts
  - Buffalo General Hospital, Department of Orthopaedics Kaleida Health, Buffalo, New York
  - Crystal Clinic, Akron, Ohio
  - The Center: Orthopaedic & Neurosurgical Care & Research, Bend, Oregon
  - Knoxville Orthopaedic Clinic, Knoxville, Tennessee
  - Scott & White Memorial Hospital, Temple, Texas
  - Aurora Advanced Healthcare, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 467/500 participants/knees enrolled;56 participants/60 knees censored = 411/440 participants/knees followed
Groups:
- Triathlon® CR Total Knee System: Participants who received the Triathlon® CR Total Knee System can have one or both knees replaced. If both knees were replaced, but only one knee completed the study, the participant is counted as having completed.
Period: Overall Study
Arm/Group | Triathlon® CR Total Knee System
Started | 411
Completed | 298 (Completed/Not completed counts are based on participant status at the 2yr primary outcome interval.)
Not Completed | 113
Not completed — Death | 3
Not completed — Revision/ Removal of Study Implant | 3
Not completed — Lost to Follow-up | 8
Not completed — Withdrawal by Subject | 24
Not completed — Investigative Site Terminated | 61
Not completed — Intercurrent Illness | 2
Not completed — 2yr ROM Data Not Evaluable | 12

BASELINE CHARACTERISTICS:
Groups:
- Triathlon® CR Total Knee System: Participants who received the Triathlon® CR Total Knee System and were not censored from analysis.
Arm/Group | Triathlon® CR Total Knee System
Number analyzed (Participants) | 411
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 239
  Male | 172
Region of Enrollment [Number; unit: participants]
  United States | 411

OUTCOME MEASURES:

1. Primary Outcome: Active Range of Motion
Time Frame: 2 Years
Population: Participants/knees with available data.
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: knees
Groups:
- Triathlon® CR Total Knee System: Non-censored participants/knees who received the Triathlon® CR Total Knee System
Arm/Group | Triathlon® CR Total Knee System
Number analyzed (Participants) | 298
Number analyzed (knees) | 317
Degrees | 119.2 (10.66)

2. Secondary Outcome: Change in Knee Society Score (KSS) Over Time
Description: The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, ROM and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: preoperative, 1, 2, and 5 years
Population: Participants/knees with available data. Overall number of participants and units analyzed is based upon the preoperative population.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: knees
Arm/Group | Triathlon® CR Total Knee System
Number analyzed (Participants) | 410
Number analyzed (knees) | 439
units on a scale
  Pain/Motion Mean Preoperative Score: number analyzed (Participants) | 387
  Pain/Motion Mean Preoperative Score: number analyzed (knees) | 414
  Pain/Motion Mean Preoperative Score | 37.39 (13.80)
  Pain/Motion Mean 1 Year Score: number analyzed (Participants) | 340
  Pain/Motion Mean 1 Year Score: number analyzed (knees) | 364
  Pain/Motion Mean 1 Year Score | 92.12 (10.13)
  Pain/Motion Mean 2 Year Score: number analyzed (Participants) | 280
  Pain/Motion Mean 2 Year Score: number analyzed (knees) | 298
  Pain/Motion Mean 2 Year Score | 93.83 (7.93)
  Pain/Motion Mean 5 Year Score: number analyzed (Participants) | 185
  Pain/Motion Mean 5 Year Score: number analyzed (knees) | 190
  Pain/Motion Mean 5 Year Score | 94.86 (8.48)
  Function Mean Preoperative Score | 53.34 (17.46)
  Function Mean 1 Year Score: number analyzed (Participants) | 359
  Function Mean 1 Year Score: number analyzed (knees) | 385
  Function Mean 1 Year Score | 86.04 (17.40)
  Function Mean 2 Year Score: number analyzed (Participants) | 290
  Function Mean 2 Year Score: number analyzed (knees) | 309
  Function Mean 2 Year Score | 86.08 (17.98)
  Function Mean 5 Year Score: number analyzed (Participants) | 198
  Function Mean 5 Year Score: number analyzed (knees) | 203
  Function Mean 5 Year Score | 85.49 (19.62)
Statistical Analysis 1: Comparison: Triathlon® CR Total Knee System; Change from pre-op to 1 year, 2 year and 5 year; Test type: Superiority or Other; p < 0.0001, Sign test

3. Secondary Outcome: Active Flexion, Passive Flexion, Active Extension, and Passive Extension Range of Motion (ROM)
Description: Knee range of motion is measured by the number of degrees flexion and extension observed. Active motion is the number of degrees that a participant can extend and flex their knee independently. Passive motion is the number of degrees that an examiner is able to extend and flex the knee without the assistance of the participant. The Knee Society Score range of motion utilized for this study defines the range from 0 degrees of extension to 125 degrees of flexion.
Time Frame: 1, 2, and 5 years
Population: Participants/knees with available data. Overall number of participants and units analyzed is based upon preoperative population.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: knees
Arm/Group | Triathlon® CR Total Knee System
Number analyzed (Participants) | 360
Number analyzed (knees) | 386
degrees
  Active Flexion 1 Year | 118.47 (10.59)
  Active Flexion 2 Years: number analyzed (Participants) | 298
  Active Flexion 2 Years: number analyzed (knees) | 317
  Active Flexion 2 Years | 119.53 (10.26)
  Active Flexion 5 Years: number analyzed (Participants) | 196
  Active Flexion 5 Years: number analyzed (knees) | 201
  Active Flexion 5 Years | 120.74 (9.00)
  Active Extension 1 Year | 0.37 (1.66)
  Active Extension 2 Years: number analyzed (Participants) | 298
  Active Extension 2 Years: number analyzed (knees) | 317
  Active Extension 2 Years | 0.28 (1.71)
  Active Extension 5 Years: number analyzed (Participants) | 196
  Active Extension 5 Years: number analyzed (knees) | 201
  Active Extension 5 Years | 0.26 (1.49)
  Passive Flexion 1 Year: number analyzed (Participants) | 359
  Passive Flexion 1 Year: number analyzed (knees) | 385
  Passive Flexion 1 Year | 121.55 (10.43)
  Passive Flexion 2 Years: number analyzed (Participants) | 293
  Passive Flexion 2 Years: number analyzed (knees) | 312
  Passive Flexion 2 Years | 122.89 (10.39)
  Passive Flexion 5 Years: number analyzed (Participants) | 192
  Passive Flexion 5 Years: number analyzed (knees) | 197
  Passive Flexion 5 Years | 123.41 (8.53)
  Passive Extension 1 Year: number analyzed (Participants) | 359
  Passive Extension 1 Year: number analyzed (knees) | 385
  Passive Extension 1 Year | 0.19 (1.23)
  Passive Extension 2 Years: number analyzed (Participants) | 293
  Passive Extension 2 Years: number analyzed (knees) | 312
  Passive Extension 2 Years | 0.08 (0.91)
  Passive Extension 5 Years: number analyzed (Participants) | 192
  Passive Extension 5 Years: number analyzed (knees) | 197
  Passive Extension 5 Years | 0.16 (1.01)
Statistical Analysis 1: Comparison: Triathlon® CR Total Knee System; Change from pre-op to 1, 2, and 5 year; Test type: Superiority or Other; p < 0.0001, Sign test

4. Secondary Outcome: Number of Knees With Radiographic Failure Assessed Via the Knee Society Total Knee Arthroplasty Roentgenographic Score
Description: Parameters for radiographic failures will follow the guidelines that have been set by the Knee Society. The scoring system for each of the three components is determined by measuring the width of the radiolucent lines for each of the zones in millimeters for each of the three components. The total widths in millimeters are added for each zone for each of the three prostheses. The total produces a numerical score for each component. Failure is defined as a score of 10 or greater, regardless of symptoms.
Time Frame: 1, 2, and 5 years
Population: Participants/knees with available data. Overall number of participants and units analyzed is based upon the one year population.
Measure: Number; unit: Total number of knees
Units Other Than Participants: knees
Arm/Group | Triathlon® CR Total Knee System
Number analyzed (Participants) | 347
Number analyzed (knees) | 370
Total number of knees
  Radiographic Failure at 1 Year | 1
  Radiographic Failure at 2 Years: number analyzed (Participants) | 295
  Radiographic Failure at 2 Years: number analyzed (knees) | 314
  Radiographic Failure at 2 Years | 1
  Radiographic Failure at 5 Years: number analyzed (Participants) | 198
  Radiographic Failure at 5 Years: number analyzed (knees) | 203
  Radiographic Failure at 5 Years | 0

5. Secondary Outcome: Change in SF-36 Health Survey Over Time
Description: The SF-36 Health Survey is a 36 item patient completed questionnaire to measure general health and well-being. It includes a physical and mental status component score; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: preoperative, 1, 2, 3, 4, and 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: knees
Arm/Group | Triathlon® CR Total Knee System
Number analyzed (Participants) | 403
Number analyzed (knees) | 432
units on a scale
  Physical Score Preoperative | 32.54 (7.50)
  Physical Score 1 Year: number analyzed (Participants) | 356
  Physical Score 1 Year: number analyzed (knees) | 379
  Physical Score 1 Year | 47.77 (7.96)
  Physical Score 2 Years: number analyzed (Participants) | 284
  Physical Score 2 Years: number analyzed (knees) | 303
  Physical Score 2 Years | 47.48 (8.71)
  Physical Score 3 Years: number analyzed (Participants) | 258
  Physical Score 3 Years: number analyzed (knees) | 270
  Physical Score 3 Years | 46.94 (9.06)
  Physical Score 4 Years: number analyzed (Participants) | 219
  Physical Score 4 Years: number analyzed (knees) | 223
  Physical Score 4 Years | 46.22 (9.46)
  Physical score 5 Years: number analyzed (Participants) | 190
  Physical score 5 Years: number analyzed (knees) | 195
  Physical score 5 Years | 46.04 (9.57)
  Mental Score Preoperative | 52.55 (12.13)
  Mental Score 1 Year: number analyzed (Participants) | 356
  Mental Score 1 Year: number analyzed (knees) | 379
  Mental Score 1 Year | 55.60 (7.79)
  Mental Score 2 Years: number analyzed (Participants) | 284
  Mental Score 2 Years: number analyzed (knees) | 303
  Mental Score 2 Years | 55.79 (7.86)
  Mental Score 3 Years: number analyzed (Participants) | 258
  Mental Score 3 Years: number analyzed (knees) | 270
  Mental Score 3 Years | 55.53 (7.72)
  Mental Score 4 Years: number analyzed (Participants) | 219
  Mental Score 4 Years: number analyzed (knees) | 223
  Mental Score 4 Years | 54.72 (7.87)
  Mental Score 5 Years: number analyzed (Participants) | 190
  Mental Score 5 Years: number analyzed (knees) | 195
  Mental Score 5 Years | 55.65 (8.37)
Statistical Analysis 1: Comparison: Triathlon® CR Total Knee System; SF36 Physical Component Score change from preop to 1 year; Test type: Superiority or Other; p < 0.0001, Sign test
Statistical Analysis 2: Comparison: Triathlon® CR Total Knee System; SF36 Mental Component Score change from preop to 1 year; Test type: Superiority or Other; p = 0.0002, Sign test
Statistical Analysis 3: Comparison: Triathlon® CR Total Knee System; SF36 Physical Component Score change from preop to 2 years; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Triathlon® CR Total Knee System; SF36 Mental Component Score change from preop to 2 years; Test type: Superiority or Other; p = 0.0177, Sign test
Statistical Analysis 5: Comparison: Triathlon® CR Total Knee System; SF36 Physical Component Score change from preop to 3 year; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 6: Comparison: Triathlon® CR Total Knee System; SF36 Mental Component Score change from preop to 3 year; Test type: Superiority or Other; p = 0.0393, Sign test
Statistical Analysis 7: Comparison: Triathlon® CR Total Knee System; SF36 Physical Component Score change from preop to 4 year; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 8: Comparison: Triathlon® CR Total Knee System; SF36 Mental Component Score change from preop to 4 year; Test type: Superiority or Other; p = 0.4905, t-test, 2 sided
Statistical Analysis 9: Comparison: Triathlon® CR Total Knee System; SF36 Physical Component Score change from preop to 5 year; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 10: Comparison: Triathlon® CR Total Knee System; SF36 Mental Component Score change from preop to 5 year; Test type: Superiority or Other; p = 0.0037, Sign test

6. Secondary Outcome: Change in Western Ontario and McMaster Osteoarthritis Index (WOMAC) Over Time
Description: The WOMAC collects information specific to osteoarthritis outcomes. The questionnaire uses a visual analog scale for pain, measuring factors of general pain, stiffness, and physical findings. Pain is scored from 0 to 100 for each set of factors, with 0 indicating no pain and 100 indicating extreme pain. Total WOMAC scores range from 0 to 300. Lower values represent better outcomes.
Time Frame: preoperative,1, 2, 3, 4 and 5 years
Population: Participants/knees with available data. Data for the WOMAC is only available at the 2, 3, 4 and 5 year intervals in limited numbers due to typographical errors noted on earlier interval forms rendering them invalid for comparison.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: knees
Arm/Group | Triathlon® CR Total Knee System
Number analyzed (Participants) | 94
Number analyzed (knees) | 97
units on a scale
  Total WOMAC 2 Years: number analyzed (Participants) | 1
  Total WOMAC 2 Years: number analyzed (knees) | 1
  Total WOMAC 2 Years | 94.54
  Total WOMAC 3 Years: number analyzed (Participants) | 1
  Total WOMAC 3 Years: number analyzed (knees) | 1
  Total WOMAC 3 Years | 11.68
  Total WOMAC 4 Years: number analyzed (Participants) | 50
  Total WOMAC 4 Years: number analyzed (knees) | 51
  Total WOMAC 4 Years | 36.33 (48.92)
  Total WOMAC 5 Years | 26.71 (36.18)

7. Secondary Outcome: Change in Lower-Extremity Activity Scale (LEAS) Over Time
Description: The LEAS is completed by the participant to assess activity level. Activity levels were ordered in terms of intensity from 1 to 18, with 18 indicating the highest activity level.
Time Frame: preoperative, 1, 2, 3, 4, and 5 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: knees
Arm/Group | Triathlon® CR Total Knee System
Number analyzed (Participants) | 409
Number analyzed (knees) | 438
units on a scale
  LEAS Preoperative | 9.30 (2.87)
  LEAS 1 Year: number analyzed (Participants) | 356
  LEAS 1 Year: number analyzed (knees) | 380
  LEAS 1 Year | 11.22 (2.71)
  LEAS 2 Years: number analyzed (Participants) | 286
  LEAS 2 Years: number analyzed (knees) | 304
  LEAS 2 Years | 11.45 (2.91)
  LEAS 3 Years: number analyzed (Participants) | 261
  LEAS 3 Years: number analyzed (knees) | 273
  LEAS 3 Years | 11.10 (2.76)
  LEAS 4 Years: number analyzed (Participants) | 218
  LEAS 4 Years: number analyzed (knees) | 222
  LEAS 4 Years | 11.10 (2.89)
  LEAS 5 Years: number analyzed (Participants) | 196
  LEAS 5 Years: number analyzed (knees) | 201
  LEAS 5 Years | 11.44 (2.94)
Statistical Analysis 1: Comparison: Triathlon® CR Total Knee System; LEAS score change from preop to 1, 2, 3, 4, and 5 years; Test type: Superiority or Other; p < 0.0001, Sign test

8. Secondary Outcome: Patellar Subluxation, Dislocation and Fracture Rate
Description: The incidence of patellar subluxation, dislocation or fracture is reported.
Time Frame: 5 years
Population: Participants/knees with available data at 5 years.
Measure: Count of Units; unit: knees
Units Other Than Participants: knees
Arm/Group | Triathlon® CR Total Knee System
Number analyzed (Participants) | 210
Number analyzed (knees) | 215
knees
  Patellar fracture | 4
  Patellar subluxation | 0
  Patellar dislocation | 0

9. Secondary Outcome: Patient Outcome Long Term Follow-up Questionnaire Over Time
Description: Patient-reported outcome is collected using a long-term follow-up questionnaire at 6, 7, 8, 9, and 10 years postoperative for the subjects who consent to participation in the long-term follow-up study. The questionnaire consists of three yes or no questions:
  1. Do you have any pain in your knee that has the study knee replacement?
  2. Are you satisfied with the results of your study total knee replacement?
  3. Have you had any surgery on your study knee since the time of your last study required visit/contact?
Time Frame: 6, 7, 8, 9, and 10 years
Population: Participants/knees with available data. Overall number of participants and units analyzed is based upon the eight year postoperative population, as this was the largest available population between the 6-10 year postoperative intervals.
Measure: Count of Units; unit: knees
Units Other Than Participants: knees
Groups:
- Triathlon® CR Total Knee System: Non-censored participants/knees who received the Triathlon® CR Total Knee System, and consented to the long-term follow-up study.
Arm/Group | Triathlon® CR Total Knee System
Number analyzed (Participants) | 93
Number analyzed (knees) | 93
knees
  Pain in Study Knee at 6 Yr: number analyzed (Participants) | 46
  Pain in Study Knee at 6 Yr: number analyzed (knees) | 47
  Pain in Study Knee at 6 Yr | 8
  Pain in Study Knee at 7 Yr: number analyzed (Participants) | 79
  Pain in Study Knee at 7 Yr: number analyzed (knees) | 79
  Pain in Study Knee at 7 Yr | 9
  Pain in Study Knee at 8 Yr | 8
  Pain in Study Knee at 9 Yr: number analyzed (Participants) | 87
  Pain in Study Knee at 9 Yr: number analyzed (knees) | 87
  Pain in Study Knee at 9 Yr | 9
  Pain in Study Knee at 10 Yr: number analyzed (Participants) | 90
  Pain in Study Knee at 10 Yr: number analyzed (knees) | 91
  Pain in Study Knee at 10 Yr | 9
  Satisfied with Results of Knee Replacement at 6 Yr: number analyzed (Participants) | 46
  Satisfied with Results of Knee Replacement at 6 Yr: number analyzed (knees) | 47
  Satisfied with Results of Knee Replacement at 6 Yr | 47
  Satisfied with Results of Knee Replacement at 7 Yr: number analyzed (Participants) | 79
  Satisfied with Results of Knee Replacement at 7 Yr: number analyzed (knees) | 79
  Satisfied with Results of Knee Replacement at 7 Yr | 79
  Satisfied with Results of Knee Replacement at 8 Yr | 88
  Satisfied with Results of Knee Replacement at 9 Yr: number analyzed (Participants) | 87
  Satisfied with Results of Knee Replacement at 9 Yr: number analyzed (knees) | 87
  Satisfied with Results of Knee Replacement at 9 Yr | 83
  Satisfied with Results of Knee Replacement at 10Yr: number analyzed (Participants) | 90
  Satisfied with Results of Knee Replacement at 10Yr: number analyzed (knees) | 91
  Satisfied with Results of Knee Replacement at 10Yr | 89
  Absence of Surgery on Study Knee at 6 Yr: number analyzed (Participants) | 46
  Absence of Surgery on Study Knee at 6 Yr: number analyzed (knees) | 47
  Absence of Surgery on Study Knee at 6 Yr | 47
  Absence of Surgery on Study Knee at 7 Yr: number analyzed (Participants) | 79
  Absence of Surgery on Study Knee at 7 Yr: number analyzed (knees) | 79
  Absence of Surgery on Study Knee at 7 Yr | 79
  Absence of Surgery on Study Knee at 8 Yr | 93
  Absence of Surgery on Study Knee at 9 Yr: number analyzed (Participants) | 87
  Absence of Surgery on Study Knee at 9 Yr: number analyzed (knees) | 87
  Absence of Surgery on Study Knee at 9 Yr | 87
  Absence of Surgery on Study Knee at 10 Yr: number analyzed (Participants) | 90
  Absence of Surgery on Study Knee at 10 Yr: number analyzed (knees) | 91
  Absence of Surgery on Study Knee at 10 Yr | 91

10. Secondary Outcome: Implant Survivorship
Description: Implant survivorship at 10 years postoperative is determined using the Kaplan-Meier method.
Time Frame: 10 years
Population: Participants with available data.
Measure: Number; unit: percentage of knees
Units Other Than Participants: knees
Arm/Group | Triathlon® CR Total Knee System
Number analyzed (Participants) | 411
Number analyzed (knees) | 440
percentage of knees
  Kaplan-Meier estimate (based on 5-year cases) | 98.62
  Kaplan-Meier estimate (based on 10-year cases): number analyzed (Participants) | 106
  Kaplan-Meier estimate (based on 10-year cases): number analyzed (knees) | 108
  Kaplan-Meier estimate (based on 10-year cases) | 100

ADVERSE EVENTS:
Time Frame: To 10 yrs postop. Initially, all AEs reported then modified to operative-site (serious/non-serious) and serious systemic. Years 6-10 operative-site (serious/non-serious) & any AE deemed to be related or uncertain in relation to device.
Description: Censored were not included as at risk. Industry Standard AE terms not used; specific AE terms not used for all AEs. Elective procedures not included eg. non-study joint replacement/revision, rotator cuff repair, carpal tunnel release, cataract, intra-ocular & bunion procedures, total shoulder repair, laminectomy, microdiscectomy, breast reduction, cervical spine fusion & mid-foot/flat-foot surgery.
Groups:
- Operative-Site Adverse Events: Participants who received the Triathlon® CR Total Knee System and were not censored from analysis. Operative-site events are reported by knee.
- Systemic Adverse Events: Participants who received the Triathlon® CR Total Knee System and were not censored from analysis. Systemic events are reported by participant.
Arm/Group | Operative-Site Adverse Events | Systemic Adverse Events
Serious Adverse Events (participants affected / at risk) | 21/440 | 90/411
Other Adverse Events (participants affected / at risk) | 79/440 | 0/411
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Operative-Site Adverse Events (N=440) | Systemic Adverse Events (N=411)
Operative Site (Blood and lymphatic system disorders) | 1 (1) | 0/0 (0)
Systemic (Cardiac disorders) | 0/0 (0) | 22 (25)
Systemic (Eye disorders) | 0/0 (0) | 1 (1)
Systemic (Gastrointestinal disorders) | 0/0 (0) | 16 (18)
Systemic (General disorders) | 0/0 (0) | 4 (4)
Systemic (Infections and infestations) | 0 (0) | 5 (6)
Systemic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Operative-Site (Musculoskeletal and connective tissue disorders) | 13 (15) | 0/0 (0)
Systemic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/0 (0) | 19 (26)
Operative-Site (Nervous system disorders) | 2 (2) | 0/0 (0)
Systemic (Psychiatric disorders) | 0/0 (0) | 1 (1)
Systemic (Renal and urinary disorders) | 0/0 (0) | 6 (6)
Systemic (Reproductive system and breast disorders) | 0/0 (0) | 1 (1)
Operative-Site (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0/0 (0)
Systemic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Operative-Site (Vascular disorders) | 5 (5) | 0/0 (0)
Systemic (Blood and lymphatic system disorders) | 0/0 (0) | 3 (3)
Systemic (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 13 (14)
Systemic (Nervous system disorders) | 0/0 (0) | 3 (4)
Systemic (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 11 (11)
Systemic (Vascular disorders) | 0/0 (0) | 10 (10)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operative-Site Adverse Events (N=440) | Systemic Adverse Events (N=411)
Operative Site (Musculoskeletal and connective tissue disorders) | 79 (93) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each investigator shall have privileges for their own center's results at the completion of the study. These manuscripts and abstracts will be delayed until after the multi-center publication is submitted.All publications shall be submitted to the sponsor for review at least 60 days prior to submission for publication.The sponsor shall not edit or otherwise influence the publications other than to ensure that confidential information is not disclosed and that the data is accurately represented.